CLINICAL TRIAL: NCT01842516
Title: A Phase I Clinical Study, Randomized, Double-blind, Placebo-controlled, Multiple Doses, Dose Escalation Study of the Safety, Tolerability, and Population Pharmacokinetics of LCB01-0371 in Healthy Male Subjects.
Brief Title: Multiple Ascending Dose Study for LCB01-0371
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCB01-0371-12-1-02
Record Dates: First submitted 2013-04-20; First posted 2013-04-29 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
MeSH Terms: interventions — delpazolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LCB01-0371 800mg (Experimental): LCB01-0371 800mg
  Interventions: Drug: LCB01-0371 800mg
- LCB01-0371 1200mg (Experimental): LCB01-0371 1200mg
  Interventions: Drug: LCB01-0371 1200mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCB01-0371 800mg — LCB0-0371 800mg
  Other Names: LCB0-0371 800mg
  Arms: LCB01-0371 800mg
Drug: LCB01-0371 1200mg — LCB01-0371 1200mg
  Arms: LCB01-0371 1200mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Primary

* To investigate the safety and tolerability of LCB01-0371 after a multiple oral dose
* To investigate the pharmacokinetic characteristics of LCB01-0371 after a multiple oral dose in healthy male subjects
* To investigate the safety of LCB01-0371 after a multiple oral dose in healthy male subjects

DETAILED DESCRIPTION:
* To investigate the PK characteristics of LCB01-0371 after a multiple oral dose
* To investigate the safety and tolerability of LCB01-0371 after a multiple oral dose

ELIGIBILITY:
Inclusion Criteria:

1. Health Male between 20 and 45 years of age at the time of screening and a subject with body mass index (BMI) between 19 and 27
2. Medically healthy with no clinically significant screening results through Physical examination, x-ray, 12 lead ECG, Laboratory test
3. Able to donate blood during study period and follow visit.
4. Agree to continue to use a reliable method of birth control until 60 days after study completion.
5. Capable of giving written informed consent and Able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

1. History of liver, kidney, respiratory, musculoskeletal, endocrinologic, neuropsychiatric, hemato-oncologic, or cardiovascular problem(s).
2. History of gastrointestinal problem which is affect to absorption within 6 months from screening
3. History of hypersensitivity or clinically significant adverse drug reaction(s) to the LCB01-0371, same class of the study drugs (linezolid), or other drugs including aspirin and antibiotics.
4. History drug abuse or positive result of urine drug screening test for amphetamine, methamphetamine, barbiturate, cocaine, opiate, benzodiazepine, cannabinoid, methadone, etc.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 7 days

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of LCB01-0371 | Up to 7 days
Peak Plasma Concentration (Cmax) of LCB01-0371 | Up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, MD, PhD., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho YS, Lim HS, Cho YL, Nam HS, Bae KS. Multiple-dose Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral LCB01-0371 in Healthy Male Volunteers. Clin Ther. 2018 Dec;40(12):2050-2064. doi: 10.1016/j.clinthera.2018.10.007. Epub 2018 Nov 10. PMID 30420289